CLINICAL TRIAL: NCT06518135
Title: Axillary Sentinel Lymph Node Biopsy After Neoadjuvant Chemotherapy in Patients With Initial cN1 Breast Cancer: a Prospective, Multicenter, Single Arm, Real World Study
Brief Title: Axillary Sentinel Lymph Node Biopsy After Neoadjuvant Chemotherapy in Patients With Initial cN1 Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2024-157
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-05

CONDITIONS: Sentinel Lymph Node Biopsy
Keywords: Axillary sentinel lymph node biopsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SLNB group: Standard sentinel lymph node biopsy group, if frozen pathology SLNs are negative, no ALND will be performed; If frozen pathological SLNs are positive, ALND should be performed directly; If the frozen pathology is false negative, it is recommended to complete ALND within 12 weeks after SLNB surgery.
  Interventions: Other: SLNB group

INTERVENTIONS:
Other: SLNB group — After the completion of neoadjuvant therapy, axillary SLNB should be performed first before breast surgery; If the frozen pathology SLNs are negative, ALND will no longer be performed; If frozen pathological SLNs are positive, ALND should be performed directly; If frozen pathology is false negative.
  Other Names: experimental group

SUMMARY:
SLNB has been recommended by domestic and foreign guidelines for patients with initial cN1 and NAC descending to ycN0. However, the best technical path is still not very clear at present, and the long-term tumor safety data is still insufficient. Therefore, it is necessary to further explore the optimal technical pathway and long-term tumor safety for SLNB in patients with initial cN1 and NAC downgrading to ycN0 in the real world.This study will evaluate the optimized technical pathway and long-term tumor safety of SLNB in patients with initial cN1 and NAC downgrading to ycN0 in real-world studies.

DETAILED DESCRIPTION:
SLNB has been recommended by domestic and foreign guidelines for patients with initial cN1 and NAC descending to ycN0. However, the best technical path is still not very clear at present, and the long-term tumor safety data is still insufficient. Therefore, it is necessary to further explore the optimal technical pathway and long-term tumor safety for SLNB in patients with initial cN1 and NAC downgrading to ycN0 in the real world.This study will evaluate the optimized technical pathway and long-term tumor safety of SLNB in patients with initial cN1 and NAC downgrading to ycN0 in real-world studies. The main endpoint of the study was axillary recurrence free survival. The secondary study endpoints were regional lymph node recurrence free survival, disease-free survival, overall survival, incidence of postoperative upper limb lymphedema, and patient quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Patients With ECOG Score 0-1 Points
2. Patients With Breast Cancer Stage cT1-3N1M0 (According to AJCC Version 7) Pathological Diagnosis of Ipsilateral Axillary Lymph Node Metastasis in Patients With Invasive Breast Cancer
3. Patients With Abnormal Axillary Lymph Nodes ≤ 3 Detected by Imaging Examination
4. Patients With Effective Neoadjuvant Therapy (CR+PR)
5. Patients With Clinical Axillary Negative ycN0 After Neoadjuvant Therapy
6. Patients Without Prior History of Ipsilateral Axillary Surgery and Radiation Therapy
7. Patients Without Previous History of Ipsilateral Breast Cancer (Including Carcinoma in Situ)
8. Patients Without Obvious Contraindications for Surgery or Radiation Therapy
9. No Other History of Malignant Tumors Within 5 Years From Enrollment in the Study
10. Patients Who Participate in Other Clinical Trials at the Same Time and Are Judged by the Researchers Not to Affect the Study Protocol Can be Enrolled Normally
11. The patient voluntarily joined this study and signed an informed consent form.

Exclusion Criteria:

1. Stage IV (metastatic) breast cancer；
2. Simultaneous double breast cancer；
3. Baseline cT4;
4. Baseline cN2-3
5. gestation
6. There are contraindications for SLNB;
7. Suffering from serious comorbidities or other comorbidities that may interfere with the planned treatment, or any other circumstances in which the researcher deems the patient unsuitable to participate in this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients with positive initial cT1-3N1 axillary lymph nodes
Sampling Method: Non-Probability Sample
Enrollment: 508 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Axillary recurrence-free survival | 5th year after surgery
  The time from surgery to axillary recurrence or last follow-up

SECONDARY OUTCOMES:
regional lymph node recurrence-free survival | 5th year after surgery
  The time from surgery to the occurrence of regional lymph node recurrence, metastasis, or last follow-up
Disease-free survival | 5th year after surgery
  The time from surgery to the occurrence of recurrence, metastasis, or last follow-up
Overall survival | 5th year after surgery
  The time from surgery to patient death or last follow-up
The incidence of postoperative upper limb lymphedema | 5th year after surgery
  By using the circumference method, the styloid process of the ulna is taken as the starting point, with an interval of 10cm and measured up to 40cm. The circumference is measured, and the volume of the affected limb is ≥ 10% or>200ml.
EORTC-QLQ-C30 V3 rating | 5th year after surgery
  The EORTC-QLQ-C30 V3 is the core scale of the quality of life measurement system developed by the European Organization for Research and Treatment of Cancer (EORTC) for cancer patients.
  The scale consists of 30 items, including 5 functional scales (physical function, role function, cognitive function, emotional function, social function), 3 symptom scales (fatigue, pain, malignant vomiting), 6 individual measurement items (swallowing difficulties, loss of appetite, sleep disorders, constipation, diarrhea, economic difficulties), and 1 patient self-assessment item (overall health status).
  The original scores for each item need to be converted into standardized scores ranging from 0 to 100 using a linear formula. The higher the score for each functional dimension, the better the functional status; The higher the score of the symptom scale and individual items, the more obvious the symptoms and the poorer the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenzhen Liu, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan cacer hospital, Henan, Henan, China